CLINICAL TRIAL: NCT07118020
Title: A Prospective Post-Market Study of Tutopatch in Craniotomy
Brief Title: Post Market Study of Tutopatch In Craniotomy
Status: Enrolling by invitation | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: RTI-2022-02
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a post market prospective, multi-center study of up to 75 participants at approximately 8 clinical study sites. The objective of the study is to evaluate safety by assessing incidence of device and/or procedure related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any age undergoing craniotomy
* Able to return for scheduled study visits
* Informed consent is able to be obtained

Exclusion Criteria:

* Life expectancy < 12 months
* Local cerebral infection
* Previous surgery at same anatomical site
* Currently enrolled in another study that would affect validity of study
* Known hypersensitivity to bovine collagen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be candidates for craniotomy due to tumor, aneurysm, trauma or other medical conditions recruited from the participating investigator's population
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-09-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Device and/or Procedure Related Adverse Events | 12 months

SECONDARY OUTCOMES:
Rate of cerebrospinal fluid leakage | 12 months
Incidence of re-operation | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Universitatsklinik fur Neurochirurgie der PMU, Salzburg, Austria
- Hospital Universitari Vali d'Hebron, Barcelona, Spain